CLINICAL TRIAL: NCT02716324
Title: Communication to Improve Shared Decision-Making in Attention-Deficit/Hyperactivity Disorder
Brief Title: Communication to Improve Shared Decision-Making in ADHD
Acronym: ADHD-Link
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15-012456
Record Dates: First submitted 2016-03-10; First posted 2016-03-23 (Estimated); Results first posted 2019-09-27 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
Keywords: Attention-Deficit/Hyperactivity Disorder; Shared-Decision Making; Care Manager; Children; Parents; Teachers
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — Case Managers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADHD Portal (Active Comparator): In this arm, the ADHD Portal was used alone as an electronic communication tool.The ADHD portal is considered standard of care at our institution for communicating information between clinicians, teachers, and parents.
  Interventions: Other: ADHD Portal
- ADHD Portal plus Care Manager (CM) (Experimental): In this arm, the ADHD Portal was combined with the CM. Clinicians, teachers, and parents used the ADHD Portal as standard of care. In addition, clinicians, teachers, parents, and any external mental health providers interacted with a CM, who had access to information contained in the ADHD Portal.
  Interventions: Behavioral: Care Manager CM); Other: ADHD Portal

INTERVENTIONS:
Behavioral: Care Manager CM) — The CM was an individual responsible for communicating and coordinating ADHD care. The CM established rapport with families and communicated with them every 3 months or more frequently if needed to assess treatment use, identify new concerns, and help problem-solve. The CM also communicated with the patient's ADHD care team (pediatrician, teacher, mental health providers) to clarify family goals, communicate information, and coordinate treatment.
  Arms: ADHD Portal plus Care Manager (CM)
Other: ADHD Portal — The ADHD portal was a web-based platform that permits access to parts of the hospital's electronic health record. The portal permits (1) capture and sharing of patient and family treatment preferences and goals, (2) monitoring of ADHD symptoms, treatment receipt, and side effects, and (3) assessing goal attainment. The system prompts for completion of periodic check-in surveys (bi-weekly to 3 months) with parents and teachers. Within the portal, preferences and goals for ADHD treatment were measured using the ADHD Preference Goal Instrument (PGI) (Fiks et al., 2012). Parents were encouraged to consult with their children when completing the tool.

SUMMARY:
The purpose of this study was to explore whether using an online patient portal plus a Care Manager is more effective than using an online portal alone in managing care for children with ADHD. Doctors at The Children's Hospital of Philadelphia currently use the online patient portal to help gather information from parents and teachers on ADHD symptoms, treatment, and medication side effects. The Care Manager is a person who meets with participants during the study to discuss their child's ADHD care. The Care Manager communicates with the child's doctor and teacher to communicate a parent's goals and preferences for their child's ADHD care.

DETAILED DESCRIPTION:
Fragmentation in health care and poor communication across systems adversely impact engagement and adherence to treatment by children with ADHD and their families. Fragmentation of services for ADHD impairs communication and collaboration between families and primary care providers, mental health providers, and educators, and leads to suboptimal outcomes for children. Prior studies have documented that little communication and coordination exist among providers across different systems despite calls for better system integration.

Fragmentation in communication between providers has the potential to impair shared decision-making. To promote shared decision-making, we developed an electronic health record (EHR)-linked portal to collect information from parents, teachers and clinicians on children's ADHD symptoms and treatment-related preferences and goals. This has become standard of care at our institution. We also developed and pilot tested a ADHD Care Manager intervention which will be employed in this comparative effectiveness study.

303 participants were recruited from 11 primary care pediatric practices. Participants were randomly assigned to either the EHR portal alone, or the EHR portal plus a Care Manager. For those assigned to the EHR portal plus Care Manager, the Care Manager met with families at the beginning of the study to confirm their treatment preferences and goals, provide additional education on ADHD treatment, and distribute handouts on common concerns among ADHD patients and families. The Care Manager contacted families every 3 months or more frequently if needed by phone, email, or in-person to assess treatment use, identify new concerns, and assist families with problem-solving. The Care Manager also communicated with primary care clinicians, mental health providers, and teachers to clarify family treatment preferences and goals and address emerging treatment issues. Participants completed surveys that assessed ADHD symptoms, goal attainment, patient-reported outcomes, patient and family engagement, and treatment initiation and adherence.

ELIGIBILITY:
Inclusion Criteria:

* Aged 5 through12 years old
* Receiving Attention-Deficit/Hyperactivity Disorder (ADHD) treatment from participating practices
* ADHD or Attention Deficit Disorder (ADD) diagnosis code, International Classification of Diseases (ICD) code ICD-10-CM F90.9 or F90.0, listed in the problem list or recorded at an ambulatory visit in the past year.
* Parental/guardian permission (informed consent) and if appropriate, child assent.

Exclusion Criteria:

* Autism spectrum disorder, ICD-10-CM F84.0
* Conduct disorder, ICD-10-CM F91.1
* Psychosis, ICD-10-CM F29
* Bipolar disorder, ICD-10-CM F31.9
* Suicide attempt, ICD-10-CM T14.91, or suicide ideation, ICD-10-CM R45.85
* Children and/or their parents/caregivers non-English speaking

Ages: 5 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 303 (Actual)
Dates: Start 2016-03-10 (Actual); Primary Completion 2018-05-09 (Actual); Study Completion 2018-10-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Guevara, MD MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete, cleaned, and de-identified dataset will be made available to the Patient-Centered Outcomes Research Institute (PCORI) and other investigators after all analyses have been conducted and within nine months of the end of the final year of funding. To obtain this data set, other investigators may contact the study PI who will provide a data sharing agreement. The data sharing agreement will permit the data set to be shared once an Institutional Review Board (IRB) protocol has been approved at the investigators' home institution and the investigators have signed a pledge to not attempt to identify individual study subjects. The data set will be made available electronically or via a secure file transfer protocol (FTP) site.
Supporting Information: Study Protocol
Time Frame: July 14, 2020
Access Criteria: Contact PI

REFERENCES:
- [Background] Guevara JP, Rothbard A, Shera D, Zhao H, Forrest CB, Kelleher K, Schwarz D. Correlates of behavioral care management strategies used by primary care pediatric providers. Ambul Pediatr. 2007 Mar-Apr;7(2):160-6. doi: 10.1016/j.ambp.2006.12.006. PMID 17368411
- [Background] Forrest CB, Glade GB, Baker AE, Bocian AB, Kang M, Starfield B. The pediatric primary-specialty care interface: how pediatricians refer children and adolescents to specialty care. Arch Pediatr Adolesc Med. 1999 Jul;153(7):705-14. doi: 10.1001/archpedi.153.7.705. PMID 10401803
- [Background] Homonoff EE, Maltz PF. Developing and maintaining a coordinated system of community-based services to children. Community Ment Health J. 1991 Oct;27(5):347-58. doi: 10.1007/BF00752385. PMID 1934995
- [Background] Guevara JP, Feudtner C, Romer D, Power T, Eiraldi R, Nihtianova S, Rosales A, Ohene-Frempong J, Schwarz DF. Fragmented care for inner-city minority children with attention-deficit/hyperactivity disorder. Pediatrics. 2005 Oct;116(4):e512-7. doi: 10.1542/peds.2005-0243. PMID 16199679
- [Background] Wolraich ML, Bickman L, Lambert EW, Simmons T, Doffing MA. Intervening to improve communication between parents, teachers, and primary care providers of children with ADHD or at high risk for ADHD. J Atten Disord. 2005 Aug;9(1):354-68. doi: 10.1177/1087054705278834. PMID 16371681
- [Derived] Guevara JP, Power TJ, Bevans K, Snitzer L, Leavy S, Stewart D, Broomfield C, Shah S, Grundmeier R, Michel JJ, Berkowitz S, Blum NJ, Bryan M, Griffis H, Fiks AG. Improving Care Management in Attention-Deficit/Hyperactivity Disorder: An RCT. Pediatrics. 2021 Aug;148(2):e2020031518. doi: 10.1542/peds.2020-031518. Epub 2021 Jul 19. PMID 34281997

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 3/2016-7/2017, primary care clinicians at participating pediatric practices nominated eligible patients for recruitment. Eligible patients were contacted by phone and then underwent in-person informed consent. Participants were stratified by practice, age group (5-7 or 8-12 years old), and sex and randomized 1:1 to the two study arms.
Pre-assignment Details: Eligible participants were excluded prior to enrollment if they had history of suicide, bipolar disorder, schizophrenia, autism, or conduct disorder.
Groups:
- ADHD Portal: In this arm, the ADHD Portal will be used alone as an electronic communication tool.The ADHD portal is considered standard of care at our institution for communicating information between clinicians, teachers, and parents.
  ADHD Portal: The ADHD portal is a web-based platform that permits access to parts of the hospital's electronic health record. The portal permits (1) capture and sharing of patient and family treatment preferences and goals, (2) monitoring of ADHD symptoms, treatment receipt, and side effects, and (3) assessing goal attainment. The system prompts for completion of periodic check-in surveys (bi-weekly to 3 months) with parents and teachers. Within the portal, preferences and goals for ADHD treatment are measured using the ADHD Preference Goal Instrument (PGI) (Fiks et al., 2012). Parents are encouraged to consult with their children when completing the tool.
- ADHD Portal Plus Care Manager: In this arm, the ADHD Portal is combined with the Care Manager. Clinicians, teachers, and parents will use the ADHD Portal. Clinicians, teachers, parents, and any external mental health providers will interact with a Care Manager, who will have access to information contained in the ADHD Portal.
  Care Manager: The CM is responsible for communicating and coordinating ADHD care. The CM communicates with families weekly-every 3 months to assess treatment use and concerns, and problem-solve. The CM communicates with their ADHD care team (pediatrician, teacher, mental health provider) to clarify goals, communicate information, and coordinate treatment.
  ADHD Portal: The ADHD portal is a web platform that permits access to parts of CHOP's electronic health record. The portal permits 1) capture, sharing of treatment preferences. 2) monitoring of ADHD symptoms, treatments, and side effects, and 3) assessing goal attainment.
Period: Overall Study
Arm/Group | ADHD Portal | ADHD Portal Plus Care Manager
Started | 149 | 154
Completed | 130 | 143
Not Completed | 19 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADHD Portal | ADHD Portal Plus Care Manager | Total
Number analyzed (Participants) | 149 | 154 | 303
Age, Categorical [Count of Participants; unit: Participants] — Population: Participants were recruited between ages five to twelve years old.
  Participants
    <=18 years | 149 | 154 | 303
    Between 18 and 65 years | 0 | 0 | 0
    >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: It was expected that the gender distribution would reflect the gender distribution of children with ADHD in the CHOP Care Network: 72% male, 28% female. The row population differs from the overall by one as a participant did not complete further measures after consenting to the study and being randomized to the ADHD Portal Plus Care Manager Arm.
  Participants
    number analyzed (Participants) | 149 | 153 | 302
    Female | 47 | 47 | 94
    Male | 102 | 106 | 208
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: The row population differs from the overall by one as a participant did not complete further measures after consenting to the study and being randomized to the ADHD Portal Plus Care Manager Arm.
  Participants
    Race/Ethnicity: number analyzed (Participants) | 149 | 153 | 302
    Race/Ethnicity: White | 58 | 62 | 120
    Race/Ethnicity: Black/African American | 69 | 70 | 139
    Race/Ethnicity: Hispanic | 7 | 8 | 15
    Race/Ethnicity: Other | 15 | 13 | 28
Region of Enrollment [Number; unit: participants]
  United States | 149 | 154 | 303
Baseline Vanderbilt Parent Rating Scale Scores [Mean (Standard Deviation); unit: Vanderbilt Parent Rating Scale Score] — Population: The VPRS measures ADHD symptoms and is scaled on a 4-point Likert rating ("never" to "very often"). The scale includes 18 ADHD symptom items with total scores ranges from 0-54. Row differs from overall because of missing data.
  Vanderbilt Parent Rating Scale Score
    number analyzed (Participants) | 148 | 152 | 300
    (all) | 32.6 (11.8) | 31.3 (10.8) | 31.9 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: Change in Vanderbilt Parent Rating Scales (VPRS)
Description: The VPRS is a public domain tool that consists of forms completed by the child's parent and includes 18 items corresponding to the DSM-5 ADHD symptom criteria, 8 performance items, and 12 items assessing side effects. The VPRS items are scaled on a 4-point Likert rating ("never" to "very often"), and the scales used in this study were restricted to the 18 ADHD symptom items. Total scores were used to measure ADHD Symptoms. Higher scores indicated worse outcome. VPRS were measured at baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4). The time range given for Visit 4 reflects the time range counted as a single value. The VPRS measures ADHD symptoms and is scaled on a 4-point Likert rating ("never" to "very often"). The scale includes 18 ADHD symptom items with total scores ranges from 0-54.
Time Frame: Baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4)
Population: Row differs from the overall number due to missing data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ADHD Portal | ADHD Portal Plus Care Manager
Number analyzed (Participants) | 149 | 154
score on a scale
  Visit 1: number analyzed (Participants) | 148 | 152
  Visit 1 | 32.6 (11.8) | 31.3 (10.8)
  Visit 2: number analyzed (Participants) | 123 | 137
  Visit 2 | 28.7 (12.2) | 29.0 (11.4)
  Visit 3: number analyzed (Participants) | 109 | 131
  Visit 3 | 28.1 (12.1) | 26.3 (11.6)
  Visit 4: number analyzed (Participants) | 130 | 143
  Visit 4 | 27.2 (12.1) | 25.7 (11.1)
Statistical Analysis 1: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed VPRS scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. We examined intervention X time interaction term for statistical significance; Test type: Superiority; p = .871, GLS random-effects model; Beta Coefficient = 0.001, 95% CI 2-sided [-0.010 to 0.012]

2. Secondary Outcome: Mean Goal Attainment Scale (GAS) Score by Timepoint
Description: The GAS is a 5-point likert scale that assesses the degree to which parents' goals (obtained from the ADHD Preferences and Goals Instrument) are attained from none to completely. The GAS response categories are ordered from 0 ("no change") to 6 ("goal completely met"). Higher scores indicate greater goal attainment. The GAS was measured at baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4). The time range given for Visit 4 reflects the time range counted as a single value.
Time Frame: Baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4)
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | ADHD Portal | ADHD Portal Plus Care Manager
Number analyzed (Participants) | 114 | 127
Units on a scale
  Visit 2 | 2.92 (1.82) | 2.67 (1.68)
  Visit 3 | 2.93 (1.89) | 3.01 (1.68)
  Visit 4 | 3.03 (1.66) | 2.86 (1.75)
Statistical Analysis 1: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed GAS scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. We examined intervention X time interaction term for statistical significance; Test type: Superiority; p = 0.499, Random effects model; Beta coefficient = 0.001, 95% CI 2-sided [-0.002 to 0.004]

3. Secondary Outcome: Treatment Initiation and Use of Services
Description: Using responses from the Services Assessment for Children and Adolescents (SACA), a well-validated client-reported tool and provides information on any mental health services use, ambulatory services use, and inpatient service use, we determined (yes/no) whether participants ever received educational services, mental health services, or medications for ADHD. Parents reported whether their children used services ever or within the last nine months. Treatment initiation was measured by use of services ever. Categorizations include any service use, ambulatory service use (any community mental health or outpatient clinic, private professional, or in-home provider), and overnight stay (psychiatric or medical unit, residential treatment center, group home, or foster home). The time range of 9-12 given for Visit 4 reflects the time range counted as a single value.
Time Frame: 9-12 months (Visit 4)
Population: Numbers may not add to column totals due to missing data. Values and percentages for Ambulatory and Overnight services do not add up to the over n listed for the column due to missing data and logic structure of the Service Assessment for Children and Adolescents (SACA).
Measure: Count of Participants; unit: Participants
Arm/Group | ADHD Portal | ADHD Portal Plus Care Manager
Number analyzed (Participants) | 119 | 137
Participants
  Use of any services (Ever) : Yes: Yes | 79 | 88
  Use of any services (Ever) : Yes: No | 40 | 49
  Use of ambulatory services (Ever) : Yes: number analyzed (Participants) | 119 | 136
  Use of ambulatory services (Ever) : Yes: Yes | 77 | 87
  Use of ambulatory services (Ever) : Yes: No | 42 | 49
  Overnight Stay for Services (Ever) : Yes: number analyzed (Participants) | 97 | 124
  Overnight Stay for Services (Ever) : Yes: Yes | 5 | 6
  Overnight Stay for Services (Ever) : Yes: No | 92 | 118
Statistical Analysis 1: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Differences in proportions between the two groups in use of any services were assessed using the Chi-square Test; Test type: Superiority; p = 0.718, Chi-squared
Statistical Analysis 2: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Differences in proportions between the two groups in use of ambulatory mental health services were assessed using the Chi-square Test; Test type: Superiority; p = 0.903, Chi-squared
Statistical Analysis 3: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Differences in proportions between the two groups in use of any inpatient mental health services were assessed using the Chi-square Test; Test type: Superiority; p = 0.915, Chi-squared

4. Secondary Outcome: Treatment Adherence and Use of Services
Description: Using responses from the Services Assessment for Children and Adolescents (SACA), a well-validated client-reported tool and provides information on any mental health services use, ambulatory services use, and inpatient service use, we determined (yes/no) whether participants ever received educational services, mental health services, or medications for ADHD. Parents reported whether their children used services ever or within the last nine months. Treatment adherence was measured by use of services in the past nine months. Categorizations include any service use, ambulatory service use (any community mental health or outpatient clinic, private professional, or in-home provider), and overnight stay (psychiatric or medical unit, residential treatment center, group home, or foster home). The time range of 9-12 given for Visit 4 reflects the time range counted as a single value.
Time Frame: 9-12 months (Visit 4)
Population: Rows may differ from overall umber analyzed due to missing data. Values and percentages for Ambulatory and Overnight services do not add up to the over n listed for the column due to missing data and logic structure of the Service Assessment for Children and Adolescents (SACA).
Measure: Count of Participants; unit: Participants
Arm/Group | ADHD Portal | ADHD Portal Plus Care Manager
Number analyzed (Participants) | 67 | 80
Participants
  Use of any service (Past 9 months): Yes | 48 | 51
  Use of any service (Past 9 months): No | 19 | 29
  Use of ambulatory services (Past 9 months): number analyzed (Participants) | 65 | 79
  Use of ambulatory services (Past 9 months): Yes | 47 | 50
  Use of ambulatory services (Past 9 months): No | 18 | 29
  Overnight Stay for Services (Ever): number analyzed (Participants) | 4 | 6
  Overnight Stay for Services (Ever): Yes | 1 | 2
  Overnight Stay for Services (Ever): No | 3 | 4
Statistical Analysis 1: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Differences in proportions between the two groups in use of any mental health services during the study period were assessed using the Chi-square Test; Test type: Superiority; p = 0.310, Chi-squared
Statistical Analysis 2: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Differences in proportions between the two groups in use of ambulatory mental health services during the study period were assessed using the Chi-square Test; Test type: Superiority; p = 0.251, Chi-squared
Statistical Analysis 3: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Differences in proportions between the two groups in use of inpatient mental health services during the study period were assessed using the Chi-square Test; Test type: Superiority; p = 1.00, Chi-squared

5. Secondary Outcome: School Performance
Description: School Performance is a 5-item domain (minimum score=1, maximum score=5 on a 5 point Likert scale) of the of 30-item Child- (age 8-12) and 17-item Parent Patient Reported Outcomes Scores (PROS). The minimum total score for the School Performance domain is 5 and the maximum total score is 25 (total scores are not shown below). Values in the table below are reported as mean scores at each time point and therefore fall between the minimum score of 1 and maximum score of 5. Higher scores indicate better outcomes. Parent-reported PRO and child-reported PRO measures were averaged for each domain for each time point. School performance PRO scores were measured at baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4). The time range given for Visit 4 reflects the time range counted as a single value.
Time Frame: Baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4)
Population: Row values may differ from overall values due to missing data and due to child measures being completed only by children 8-12 years old.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | ADHD Portal | ADHD Portal Plus Care Manager
Number analyzed (Participants) | 148 | 150
Score on a scale
  Parent PROS : Visit 1 | 2.82 (1.00) | 2.77 (0.80)
  Parent PROS : Visit 2: number analyzed (Participants) | 114 | 125
  Parent PROS : Visit 2 | 3.00 (1.01) | 2.91 (0.80)
  Parent PROS : Visit 3: number analyzed (Participants) | 102 | 120
  Parent PROS : Visit 3 | 3.03 (0.89) | 3.04 (0.92)
  Parent PROS : Visit 4: number analyzed (Participants) | 123 | 128
  Parent PROS : Visit 4 | 3.08 (0.96) | 3.03 (0.90)
  Child PROS : Visit 1: number analyzed (Participants) | 121 | 122
  Child PROS : Visit 1 | 3.53 (0.77) | 3.42 (0.79)
  Child PROS : Visit 2: number analyzed (Participants) | 96 | 95
  Child PROS : Visit 2 | 3.22 (0.93) | 3.30 (0.81)
  Child PROS : Visit 3: number analyzed (Participants) | 81 | 100
  Child PROS : Visit 3 | 3.29 (0.85) | 3.27 (0.77)
  Child PROS : Visit 4: number analyzed (Participants) | 100 | 98
  Child PROS : Visit 4 | 3.23 (0.83) | 3.41 (0.86)
Statistical Analysis 1: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed Parent-reported PRO School Performance Scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. we examined intervention X time interaction term for statistical significance; Test type: Superiority; p = 0.662, Random effects model; Beta coefficient = 0.000, 95% CI 2-sided [-0.001 to 0.001]
Statistical Analysis 2: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed Child PRO School Performance Scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. we examined intervention X time interaction term for statistical significance; Test type: Superiority; p = 0.075, Random effects model; Beta coefficient = 0.001, 95% CI 2-sided [0.000 to 0.002]

6. Secondary Outcome: Student Engagement
Description: Student Engagement is a 4-item domain (minimum score=1, maximum score=5 on a 5 point Likert scale) of the of 30-item Child- (age 8-12) and 17-item Parent Patient Reported Outcomes Scores (PROS). The minimum total score for the Student Engagement domain is 4 and the maximum total score is 20 (total scores are not shown below). Values in the table below are reported as means at each time point and therefore fall between the minimum score of 1 and maximum score of 5. Higher scores indicate better outcomes. Parent-reported PRO and child-reported PRO measures were averaged for each domain for each time point. Student Engagement PRO scores were measured at baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4). The time range given for Visit 4 reflects the time range counted as a single value.
Time Frame: Baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | ADHD Portal | ADHD Portal Plus Care Manager
Number analyzed (Participants) | 148 | 152
Score on a scale
  Parent PROS : Visit 1 | 2.98 (0.79) | 2.93 (0.80)
  Parent PROS : Visit 2: number analyzed (Participants) | 124 | 132
  Parent PROS : Visit 2 | 3.18 (0.85) | 3.08 (0.80)
  Parent PROS : Visit 3: number analyzed (Participants) | 105 | 126
  Parent PROS : Visit 3 | 3.18 (0.78) | 3.09 (0.70)
  Parent PROS : Visit 4: number analyzed (Participants) | 123 | 133
  Parent PROS : Visit 4 | 3.24 (0.82) | 3.13 (0.80)
  Child PROS : Visit 1: number analyzed (Participants) | 121 | 122
  Child PROS : Visit 1 | 3.11 (0.82) | 3.04 (0.80)
  Child PROS : Visit 2: number analyzed (Participants) | 94 | 95
  Child PROS : Visit 2 | 3.09 (0.09) | 3.06 (0.73)
  Child PROS : Visit 3: number analyzed (Participants) | 81 | 99
  Child PROS : Visit 3 | 3.15 (0.94) | 3.01 (0.78)
  Child PROS : Visit 4: number analyzed (Participants) | 99 | 100
  Child PROS : Visit 4 | 3.08 (0.83) | 2.95 (0.79)
Statistical Analysis 1: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed Parent-reported PRO Student Engagement Scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. we examined intervention X time interaction term for statistical significance; Test type: Superiority; p = 0.707, Random effects model; Beta coefficient = 0.000, 95% CI 2-sided [-0.001 to 0.001]
Statistical Analysis 2: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed Child PRO Student Engagement Scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. we examined intervention X time interaction term for statistical significance; Test type: Superiority; p = 0.735, Random effects model; Beta coefficient = 0.000, 95% CI 2-sided [-0.001 to 0.001]

7. Secondary Outcome: Teacher Connectedness
Description: Teacher Connectedness is a 9-item domain (minimum=1, maximum=5 on a 5 point Likert scale) of the of 30-item Child- (age 8-12) and 17-item Parent Patient Reported Outcomes Scores (PROS). The minimum total score for the Teacher Connectedness domain is 9 and the maximum total score is 45 (total scores not shown below). Values in the table below are reported as means at each time point and therefore fall between the minimum score of 1 and maximum score of 5. Higher scores indicate better outcomes. Parent-reported PRO and child-reported PRO measures were averaged for each domain for each time point. Teacher Connectedness PRO scores were measured at baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4). The time range given for Visit 4 reflects the time range counted as a single value.
Time Frame: Baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4)
Population: Row values may differ from overall number analyzed due to missing data.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | ADHD Portal | ADHD Portal Plus Care Manager
Number analyzed (Participants) | 120 | 121
Score on a scale
  Child PROS : Visit 1 | 3.81 (0.80) | 3.75 (0.76)
  Child PROS : Visit 2: number analyzed (Participants) | 90 | 92
  Child PROS : Visit 2 | 3.85 (0.76) | 3.82 (0.77)
  Child PROS : Visit 3: number analyzed (Participants) | 79 | 94
  Child PROS : Visit 3 | 3.86 (0.86) | 3.77 (0.83)
  Child PROS : Visit 4: number analyzed (Participants) | 97 | 94
  Child PROS : Visit 4 | 3.75 (0.87) | 3.72 (0.84)
Statistical Analysis 1: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed Child PRO Teacher Connectedness Scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. we examined intervention X time interaction term for statistical significance; Test type: Superiority; p = 0.735, Random effects model — Random effects models regressed Child Patient Reported Outcomes Teacher Connectedness Scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. The threshold for statistical significance was p<0.05; Beta coefficient = 0.000, 95% CI 2-sided [-0.001 to 0.001]

8. Secondary Outcome: Peer Relationships
Description: Peer Relationships is a 6-item domain (minimum=1, maximum=5, on a 5 point Likert scale) of the of 30-item Child- (age 8-12) and a 7-item domain (minimum=1, maximum=5 on a 5 point Likert scale) of the 17-item Parent Patient Reported Outcomes Scores (PROS). The minimum total score is 6 and the maximum total score is 30 on the Child PROs. The minimum total score for the Peer Relationships domain is 7 and the maximum total score is 35 on the Parent PROs. Total scores not shown below. Values in the table below are reported as means at each time point and therefore fall between the minimum score of 1 and maximum score of 5. Parent-reported PRO and child-reported PRO measures were averaged for each domain for each time point. Higher scores indicate better outcomes. Peer Relationships PRO scores were measured at baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4). The time range given for Visit 4 reflects the time range counted as a single value.
Time Frame: Baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4)
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | ADHD Portal | ADHD Portal Plus Care Manager
Number analyzed (Participants) | 148 | 152
Score on a scale
  Parent PROS : Visit 1 | 3.56 (0.82) | 3.54 (0.74)
  Parent PROS : Visit 2: number analyzed (Participants) | 124 | 138
  Parent PROS : Visit 2 | 3.63 (0.75) | 3.56 (0.75)
  Parent PROS : Visit 3: number analyzed (Participants) | 110 | 129
  Parent PROS : Visit 3 | 3.61 (0.79) | 3.63 (0.74)
  Parent PROS : Visit 4: number analyzed (Participants) | 123 | 141
  Parent PROS : Visit 4 | 3.72 (0.80) | 3.66 (0.72)
  Child PROS : Visit 1: number analyzed (Participants) | 121 | 122
  Child PROS : Visit 1 | 4.03 (0.74) | 4.07 (0.71)
  Child PROS : Visit 2: number analyzed (Participants) | 97 | 100
  Child PROS : Visit 2 | 3.79 (0.75) | 3.93 (0.84)
  Child PROS : Visit 3: number analyzed (Participants) | 84 | 99
  Child PROS : Visit 3 | 3.84 (0.74) | 3.99 (0.72)
  Child PROS : Visit 4: number analyzed (Participants) | 102 | 106
  Child PROS : Visit 4 | 3.91 (0.83) | 3.94 (0.79)
Statistical Analysis 1: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed Parent-reported PRO Peer Relationship Scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. we examined intervention X time interaction term for statistical significance; Test type: Superiority; p = 0.873, Random effects model — Random effects models regressed Parent Patient Reported Outcomes Peer Relationships Scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. The threshold for statistical significance was p<0.05; Beta coefficient = 0.000, 95% CI 2-sided [-0.001 to 0.001]
Statistical Analysis 2: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed Child-reported PRO Peer Relationship Scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. we examined intervention X time interaction term for statistical significance; Test type: Superiority; p = 0.888, Random effects model — Random effects models regressed Child Patient Reported Outcomes Peer Relationships Scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. The threshold for statistical significance was p<0.05; Beta coefficient = 0.000, 95% CI 2-sided [-0.001 to 0.001]

9. Secondary Outcome: Family Relationships
Description: Family Relationships is a 6-item domain (minimum=1, maximum=5 on a 5 point Likert scale) of the 30-item Child- (age 8-12) Patient Reported Outcomes Measures of relationships with other family members over the past 4 weeks. The minimum total score for the Family Relationships domain is 6 and the maximum total score is 30 (total scores not shown below). Values in the table below are reported as means at each time point and therefore fall between the minimum score of 1 and maximum score of 5. Child-reported PRO measures were averaged for each domain for each time point. Higher scores indicate better outcomes. Family Relationships PRO scores were measured at baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4). The time range given for Visit 4 reflects the time range counted as a single value.
Time Frame: Baseline (Visit 1), 3 months (Visit 2), 6 months (Visit 3), and 9-12 months (Visit 4)
Population: Row values may differ from overall number for analysis due to missing data.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | ADHD Portal | ADHD Portal Plus Care Manager
Number analyzed (Participants) | 120 | 121
Score on a scale
  Child PROS : Visit 1 | 3.81 (0.77) | 3.82 (0.68)
  Child PROS : Visit 2: number analyzed (Participants) | 96 | 100
  Child PROS : Visit 2 | 3.83 (0.69) | 3.80 (0.65)
  Child PROS : Visit 3: number analyzed (Participants) | 85 | 102
  Child PROS : Visit 3 | 3.96 (0.67) | 3.72 (0.72)
  Child PROS : Visit 4: number analyzed (Participants) | 103 | 106
  Child PROS : Visit 4 | 3.81 (0.77) | 3.79 (076)
Statistical Analysis 1: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed Child-reported PRO Family Relationship Scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. we examined intervention X time interaction term for statistical significance; Test type: Superiority; p = 0.679, Random effects model — Random effects models regressed Child Patient Reported Outcomes Family Relationships Scores on intervention status, time (days), intervention by time, season, and clustered by doctor's office. The threshold for statistical significance was p<0.05; Beta coefficient = 0.000, 95% CI 2-sided [-0.001 to 0.001]

10. Secondary Outcome: Engagement Measure Scores
Description: The Engagement Measure is a 28-item parent self-report measure comprised of four domains: Access (5-items, total score range 5-25), Patient Family Centered Care or PFCC (6-items, total score range 6-30), Communication (3-items, total score range 3-15), and Understanding (5-items, total score range 5-25). Total scores are not reported below. Scores for each individual item and therefore the mean for each domain (means reported in the table below) ranged from 1-5 with higher scores indicating greater engagement. The time range given for Visit 4 reflects the time range counted as a single value.
Time Frame: Visit 4 (9-12 months)
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | ADHD Portal | ADHD Portal Plus Care Manager
Number analyzed (Participants) | 123 | 139
Score on a scale
  Access | 3.43 (0.7) | 3.52 (0.6)
  PFCC | 3.45 (0.7) | 3.44 (0.7)
  Communication | 2.50 (1.1) | 2.64 (1.0)
  Understanding | 2.89 (0.8) | 3.02 (0.8)
Statistical Analysis 1: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed Access Engagement Scores Scores on intervention status adjusted for season and clustered by doctor's office; Test type: Superiority; p = 0.495, Random effects model; Beta coefficient = 0.074, 95% CI 2-sided [-0.164 to 0.311]
Statistical Analysis 2: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed Patient Family Centered Care Engagement Scores Scores on intervention status adjusted for season and clustered by doctor's office; Test type: Superiority; p = 0.885, Random effects model; Beta coefficient = -0.013, 95% CI 2-sided [-0.217 to 0.191]
Statistical Analysis 3: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed Communication Engagement Scores Scores on intervention status adjusted for season and clustered by doctor's office; Test type: Superiority; p = 0.527, Random effects model; Beta coefficient = 0.073, 95% CI 2-sided [-0.182 to 0.328]
Statistical Analysis 4: Comparison: ADHD Portal vs ADHD Portal Plus Care Manager; Random effects models regressed Understanding Engagement Scores Scores on intervention status adjusted for season and clustered by doctor's office; Test type: Superiority; p = 0.285, Random effects model; Beta coefficient = 0.136, 95% CI 2-sided [-0.138 to 0.410]

ADVERSE EVENTS:
Time Frame: 9-12 months
Description: Since the study procedures were not greater than minimal risk, SAEs were not expected.
Arm/Group | ADHD Portal | ADHD Portal Plus Care Manager
All-Cause Mortality (participants affected / at risk) | 0/149 | 0/154
Serious Adverse Events (participants affected / at risk) | 0/149 | 0/154
Other Adverse Events (participants affected / at risk) | 0/149 | 0/154

LIMITATIONS AND CAVEATS:
Study was conducted within a single integrated health care system in the Philadelphia metropolitan area and results may not be generalizable to other health systems or geographic areas.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-04-17): https://cdn.clinicaltrials.gov/large-docs/24/NCT02716324/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT02716324/SAP_001.pdf